CLINICAL TRIAL: NCT03366285
Title: Bonding Quality and Gene Expression of Key Molecules Involved in Stress Response in Fullterm Infants Compared to Late Preterm Infants and Preterm Infants With Early Skin to Skin Contact or Visual Contact at Age 6 to 8 Years
Brief Title: Bonding Quality and Gene Expression in Fullterm Infants Compared to Late Preterm Infants and Preterm Infants With Early Skin to Skin or Visual Contact
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Katrin Mehler, MD, University of Cologne
Other Study IDs: 17-075
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Premature Infant
Keywords: Bonding; Gene expression; Stress response; Neurodevelopment
MeSH Terms: conditions — Premature Birth; Fractures, Stress | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral white blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Fullterm infants: Quality of bonding is assessed at 6 to 8 years of age using the attachment story completion task. Infants are recruited from the local elementary school.
  Interventions: Diagnostic Test: Attachment story completion taks (ASCT)
- Moderate to late preterm infants: Bonding quality is assessed at 6 to 8 years of age using the attachment story completion task. Infants are recruited from former participants of the "trauma and depression in late preterm parents study" (TraDelPP) conducted 2010 to 2011.
  Interventions: Diagnostic Test: Attachment story completion taks (ASCT)
- Preterm infants with skin to skin contact: Bonding quality is assessed at 6 to 8 years of age using the attachment story completion task. Infants are recruited from former participants of the "delivery room skin to skin study" (deisy) who were randomized into the skin to skin contact group. The study was conducted from 2012 to 2015.
  Interventions: Diagnostic Test: Attachment story completion taks (ASCT)
- Preterm infants with visual contact: Bonding quality is assessed at 6 to 8 years of age using the attachment story completion task. Infants are recruited from former participants of the "delivery room skin to skin study" (deisy) who were randomized into the visual contact group. The study was conducted from 2012 to 2015.
  Interventions: Diagnostic Test: Attachment story completion taks (ASCT)

INTERVENTIONS:
Diagnostic Test: Attachment story completion taks (ASCT) — Bonding quality
  Other Names: Gene expression; Self-reporting questionnaires

SUMMARY:
Recent research has identified differences in the quality of mother-child interaction and gene expression of six key molecules involved in stress response and neurobehavioral development in preterm infants (born <32 weeks of gestational age) with early skin to skin contact after birth compared to infants with visual contact at six months corrected age. We hypothesize that these differences are still identifiable at the age of 6 to 8 years and that quality of bonding in preterm infants born <32 weeks of gestation differs significantly from late preterm infants and full-term infants.

DETAILED DESCRIPTION:
Quality of bonding in former preterm infants born 2012 to 2015 who participated in the "delivery room skin to skin study" (deisy), moderate to late preterm infants born 2010 to 2011 who participated in the "trauma and depression in late preterm parents study" (TraDelPP) and full-term infants at 6 to 8 years of age is assessed using the German version of the attachment story completion task (ASCT). Additionally, gene expression of six key molecules involved in stress response and neurobehavioral development (the corticotropin releasing hormone receptor 1 and 2 genes (CRHR1 and CRHR2), arginine vasopressin gene (AVP), the glucocorticoid receptor gene (NR3C1), the serotonin receptor 2A gene (HTR2A), and the serotonin transporter gene (SLC6A4)) are quantified in in mucosal epithelial cells from buccal swabs of children of all four groups. Maternal and infant co-factors such as maternal depression, perceived social support, parental stress, infant health development and behavior are assessed by self-reporting questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* first child, singleton, former participant of "deisy" or "TraDelPP" study for preterm infants, uncomplicated vaginal birth for fullterm infants

Exclusion Criteria:

* Maternal mental health problems, resuscitation after birth, malformations or severe underlying disease

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Former preterm infants and full-term infants at 6 to 8 years of age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Bonding quality | 6 to 8 years of age
  Quality of mother infant bonding is assessed with the German version of the Attachment Story Completion Task (Bretherton and Ridgeway 1990)
Gene expression | 6 to 8 years of age
  Quantification of gene expression of six key molecules involved in stress response and neurobehavioural development

SECONDARY OUTCOMES:
Maternal depression | 6 to 8 years of age
  Maternal depression is assessed with the German long form of the Center for Epidemiological Studies Depression Scale (CES-D).
Maternal perceived social support | 6 to 8 years of age
  Perceived social support is assessed with the short version of the F-SozU scale (F-SozU K-22).
Maternal parenting stress | 6 to 8 years of age
  For the assessment of parenting stress the German version of the Parenting Stress Index (PSI) is used
Infant health and development | 6 to 8 years of age
  Infant health and development are assessed by a self-reporting questionnaire and the results from compulsory pediatric medical checkups. The questionnaire for assessment of infant health and development was designed for the KIGGS study (a large German cohort study on infant´s health)
Infant behavior | 6 to 8 years of age
  For assessment of infant behavior the German version of the Child Behavior Checklist (CBCL) is used.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cologne, Medical Faculty, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trautmann-Villalba P, Heine E, Kribs A, Mehler K. Does early skin-to-skin contact have a long-term effect on the emotional and behavioral development of very preterm infants? Front Psychol. 2024 Nov 11;15:1484419. doi: 10.3389/fpsyg.2024.1484419. eCollection 2024. PMID 39588126